CLINICAL TRIAL: NCT00565409
Title: A Randomized, Double-Blind Study Comparing the Safety & Efficacy of Once-Weekly Etanercept 50 mg, Etanercept 25 mg, & Placebo in Combination With Methotrexate in Subjects With Active Rheumatoid Arthritis
Brief Title: Study Comparing Etanercept in Combination With Methotrexate in Subjects With Rheumatoid Arthritis
Acronym: PRESERVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0881A1-4423; B1801003
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Active Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Etanercept; Drug: Methotrexate
- 2 (Active Comparator)
  Interventions: Drug: Etanercept; Drug: Methotrexate
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: Etanercept — Subcutaneous (SC), 50 mg, once weekly for 88 weeks
  Other Names: Enbrel
  Arms: 1
Drug: Methotrexate — Oral, 15 to 25 mg (varying based on dosage the subject is receiving at the time of screening and may be increased at the discretion of the investigator through Week 28 to a maximum of 25 mg/week), once weekly for 88 weeks.
  If a subject experiences an adverse event (AE) during the study, Methotrexate may be decreased by 2.5 or 5.0 mg weekly (the minimum dose to stay in the study is 10 mg/week).
  Arms: 1
Drug: Etanercept — Subcutaneous (SC), 25 mg, once weekly from week 36 to week 88.
  Arms: 2
Drug: Methotrexate — Oral, 15 to 25 mg (varying based on dosage the subject is receiving at the time of screening and may be increased at the discretion of the investigator through Week 28 to a maximum of 25 mg/week), once weekly for 88 weeks.
  If a subject experiences an adverse event (AE) during the study, Methotrexate may be decreased by 2.5 or 5.0 mg weekly (the minimum dose to stay in the study is 10 mg/week).
  Arms: 2
Drug: Placebo — Subcutaneous (SC), once weekly from week 36 to week 88.
  Arms: 3
Drug: Methotrexate — Oral, 15 to 25 mg (varying based on dosage the subject is receiving at the time of screening and may be increased at the discretion of the investigator through Week 28 to a maximum of 25 mg/week), once weekly for 88 weeks.
  If a subject experiences an adverse event (AE) during the study, Methotrexate may be decreased by 2.5 or 5.0 mg weekly (the minimum dose to stay in the study is 10 mg/week).
  Arms: 3

SUMMARY:
To compare the efficacy of the combination of etanercept 50 mg once weekly plus methotrexate with that of methotrexate monotherapy in the treatment of rheumatoid arthritis over 88 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis.
* Currently receiving an optimal dose of oral Methotrexate (MTX)(at least 15 mg/week but no more than 25 mg/week) for the treatment of rheumatoid arthritis.
* Active rheumatoid arthritis at the time of screening.

Exclusion Criteria:

* Previous or current treatment with etanercept, other tumor necrosis factor-alpha (TNF) inhibitors, or other biologic agents.
* Concurrent treatment with any disease-modifying anti-rheumatoid drugs (DMARD), other than MTX within 28 days before baseline.
* Concurrent treatment with more than 1 non-steroid anti-inflammatory drug (NSAID) at baseline.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- Australia (7):
  - Pfizer Investigational Site, Campsie, New South Wales
  - Pfizer Investigational Site, Kogarah, New South Wales
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Heidelberg West, Victoria
  - Pfizer Investigational Site, Malvern, Victoria
  - Pfizer Investigational Site, Victoria Park
- Pfizer Investigational Site, Vienna, Austria
- Belgium (3):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Yvoir
- Pfizer Investigational Site, Santiago, Santiago Metropolitan, Chile
- Colombia (2):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Czechia (5):
  - Pfizer Investigational Site, Bruntál, Czech Republic
  - Pfizer Investigational Site, Zlín, Czech Republic
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Bruntál
  - Pfizer Investigational Site, Prague
- France (8):
  - Pfizer Investigational Site, Montpellier, France
  - Pfizer Investigational Site, Corbeil-Essonnes
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Le Mans
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Eilbek
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Würzburg
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Szombathely
- Italy (3):
  - Pfizer Investigational Site, Catania, CT
  - Pfizer Investigational Site, Orbassano, TO
  - Pfizer Investigational Site, Roma
- Mexico (6):
  - Pfizer Investigational Site, Mexico City, Mexico DF
  - Pfizer Investigational Site, Guadalajara, Mexico
  - Pfizer Investigational Site, Mérida, Yucatán
  - Pfizer Investigational Site, Mexico City
  - Pfizer Investigational Site, Monterrey
  - Pfizer Investigational Site, Querétaro
- Pfizer Investigational Site, Heerlen, Netherlands
- Poland (5):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Serbia and Montenegro (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Niska Banja
- South Korea (6):
  - Pfizer Investigational Site, Seo-gu, Daejeon
  - Pfizer Investigational Site, Namdong-gu, Incheon
  - Pfizer Investigational Site, Seoul, Korea
  - Pfizer Investigational Site, Seongdong-gu, Seoul
  - Pfizer Investigational Site, Anyang-si Gyeonggi-do
  - Pfizer Investigational Site, Seoul
- Spain (6):
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, A Coruña, La Coruña
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Seville, Sevilla
- Sweden (2):
  - Pfizer Investigational Site, Falun
  - Pfizer Investigational Site, Oskarström
- Taiwan (2):
  - Pfizer Investigational Site, Tapei City, ROC
  - Pfizer Investigational Site, Kaohsiung City
- United Kingdom (2):
  - Pfizer Investigational Site, Wigan, Lancashire
  - Pfizer Investigational Site, Dudley, West Midlands

REFERENCES:
- [Derived] Tanaka Y, Smolen JS, Jones H, Szumski A, Marshall L, Emery P. The effect of deep or sustained remission on maintenance of remission after dose reduction or withdrawal of etanercept in patients with rheumatoid arthritis. Arthritis Res Ther. 2019 Jul 5;21(1):164. doi: 10.1186/s13075-019-1937-4. PMID 31277720
- [Derived] Smolen JS, Pedersen R, Jones H, Mahgoub E, Marshall L. Impact of flare on radiographic progression after etanercept continuation, tapering or withdrawal in patients with rheumatoid arthritis. Rheumatology (Oxford). 2020 Jan 1;59(1):153-164. doi: 10.1093/rheumatology/kez224. PMID 31257453
- [Derived] Smolen JS, Szumski A, Koenig AS, Jones TV, Marshall L. Predictors of remission with etanercept-methotrexate induction therapy and loss of remission with etanercept maintenance, reduction, or withdrawal in moderately active rheumatoid arthritis: results of the PRESERVE trial. Arthritis Res Ther. 2018 Jan 16;20(1):8. doi: 10.1186/s13075-017-1484-9. PMID 29338762
- [Derived] Smolen JS, Strand V, Koenig AS, Szumski A, Kotak S, Jones TV. Discordance between patient and physician assessments of global disease activity in rheumatoid arthritis and association with work productivity. Arthritis Res Ther. 2016 May 21;18(1):114. doi: 10.1186/s13075-016-1004-3. PMID 27209012
- [Derived] Smolen JS, Nash P, Durez P, Hall S, Ilivanova E, Irazoque-Palazuelos F, Miranda P, Park MC, Pavelka K, Pedersen R, Szumski A, Hammond C, Koenig AS, Vlahos B. Maintenance, reduction, or withdrawal of etanercept after treatment with etanercept and methotrexate in patients with moderate rheumatoid arthritis (PRESERVE): a randomised controlled trial. Lancet. 2013 Mar 16;381(9870):918-29. doi: 10.1016/S0140-6736(12)61811-X. Epub 2013 Jan 17. PMID 23332236
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-4423&StudyName=Study%20Comparing%20Etanercept%20in%20Combination%20with%20Methotrexate%20in%20Subjects%20With%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1: Participants received etanercept (ETN) 50 mg subcutaneous (SC) injection plus oral MTX tablet 15 to 25 mg per week for 36 weeks.
- Etanercept 50 mg Plus MTX -Period 2: Participants who were responders received etanercept 50 mg SC injection plus oral MTX (15 to 25 mg) tablet once per week for 52 weeks. Responders defined as participants with a 28 Joint Disease Activity Score (DAS28) less than or equal to (≤) 3.2 at Week 36 and an average DAS28 less than or equal to (≤) 3.2 from Week 12 visit through Week 36.
- Etanercept 25 mg Plus MTX-Period 2: Participants who were responders received etanercept 25 mg SC injection plus oral MTX (15 to 25 mg) tablet once per week for 52 weeks. Responders defined as participants with DAS28 ≤ 3.2 at Week 36 and an average DAS28 ≤ 3.2 from Week 12 visit through Week 36.
- Placebo Plus MTX-Period 2: Participants who were responders received matched placebo plus oral MTX (15 to 25 mg) tablet once per week for 52 weeks. Responders defined as participants with DAS28 ≤ 3.2 at Week 36 and an average DAS28 ≤ 3.2 from Week 12 visit through Week 36.
Period: Period 1 Open Label
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1 | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Started | 834 | 0 | 0 | 0
Completed | 756 | 0 | 0 | 0
Not Completed | 78 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Other | 21 | 0 | 0 | 0
Not completed — Protocol Violation | 14 | 0 | 0 | 0
Not completed — Unsatisfactory Response-Efficacy | 22 | 0 | 0 | 0
Not completed — no conclusion of participation record | 1 | 0 | 0 | 0
Period: After Period 1, Prior to Period 2
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1 | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Started | 756 | 0 | 0 | 0
Completed | 604 | 0 | 0 | 0
Not Completed | 152 | 0 | 0 | 0
Not completed — did not meet criteria | 152 | 0 | 0 | 0
Period: Period 2 Double-Blind
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1 | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Started | 0 | 202 | 202 | 200
Completed | 0 | 181 | 175 | 141
Not Completed | 0 | 21 | 27 | 59
Not completed — Adverse Event | 0 | 7 | 4 | 5
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 6 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Other | 0 | 4 | 5 | 9
Not completed — Unsatisfactory Response-Efficacy | 0 | 4 | 11 | 43

BASELINE CHARACTERISTICS:
Groups:
- Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1: Participants received etanercept 50 mg subcutaneous (SC) injection plus oral MTX tablet 15 to 25 mg per week for 36 weeks.
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 834
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.36 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 694
  Male | 140

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 28 Joint Disease Activity Score (DAS28) Less Than or Equal to (≤) 3.2 at Week 88
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joint count (less than [<]20 percent [%] missing SJC or PJC was prorated), erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and Patient's General Health Visual Analog Scale (VAS). VAS is a line 0-100 millimeters (mm) in length; ranged from 0 (very well)-100mm (extremely bad). Participants placed a mark indicating their health over the previous 2-3 weeks. Higher scores indicated greater affectation due to disease activity. DAS28 ≤ 3.2 units equals (=) low disease activity.
Time Frame: Week 88
Population: Modified Intent to Treat population (mITT): all participants who took at least 1 dose of double-blind test article and had at least 1 post-randomization DAS28 evaluation
Measure: Number; unit: percentage of participants
Groups:
- Etanercept 50 mg Plus MTX -Period 2: Participants who were responders received etanercept 50 mg SC injection plus oral MTX (15 to 25 mg) tablet once per week for 52 weeks. Responders defined as participants with a 28 Joint Disease Activity Score (DAS28) ≤ 3.2 at Week 36 and an average DAS28 ≤ from Week 12 visit through Week 36.
- Etanercept 25 mg Plus MTX-Period 2: Participants who were responders received etanercept 25 mg SC injection plus oral MTX (15 to 25 mg) tablet once per week for 52 weeks. Responders defined as participants with DAS28 ≤ 3.2 at Week 36 and an average DAS28 ≤ from Week 12 visit through Week 36.
- Placebo Plus MTX-Period 2: Participants who were responders received matched placebo plus oral MTX (15 to 25 mg) tablet once per week for 52 weeks. Responders defined as participants with DAS28 ≤ 3.2 at Week 36 and an average DAS28 ≤ from Week 12 visit through Week 36.
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
percentage of participants | 82.6 | 79.1 | 42.6
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Sample size estimated based on moderate/severe rheumatoid arthritis(RA) trial. Study design included only moderate RA participants, thus a low disease activity estimate of 85% (ETN+MTX) vs 70% (MTX only) assumed, required 175 randomized participants in 3 treatments for a 90% power and Type I error of 0.05 to reject the null hypothesis of no ETN+MTX vs MTX only differences. More participants qualified for Period 2 than expected, Period 2 sample size roughly 15% larger than protocol-specified; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel(CMH) test of general association, testing treatment effect on response. P-value and Odds Ratio (OR) stratified by geographic region; Loss of efficacy (LOE) imputation defined as LOE drop-outs were treated as non-responders/all other participants had LOCF applied as primary analysis; Odds Ratio (OR) = 5.36, 95% CI 2-sided [3.2 to 9.0]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Test type: Superiority or Other; p = 0.3805, Cochran-Mantel-Haenszel — P-value from CMH test of general association, testing treatment effect on response. P-value and OR stratified by geographic region; LOE imputation defined as LOE drop-outs were treated as non-responders and all other participants had LOCF applied as primary analysis; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.7 to 2.0]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.81, 95% CI 2-sided [3.0 to 7.6]

2. Secondary Outcome: Percentage of Participants Achieving DAS28 Low Disease Activity or Remission at Baseline, Weeks 4, 8, 12, 20, 28 and 36
Description: DAS28 calculated from the number of SJC and PJC using the 28 joints count, the ESR mm/hour and and Patient's General Health VAS. VAS consisted of a line 0 to 100 mm in length; ranged from 0 (very well) to 100mm (extremely bad). Participants placed a mark indicating their health over the previous 2-3 weeks. Higher scores indicated greater affectation due to disease activity. DAS28 ≤ 3.2 units = low disease activity, DAS28 < 2.6 units = remission.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28, 36
Population: Period 1 Modified Intent to Treat population (P1 mITT): all participants who took at least 1 dose of open-label test article; N=number of participants with evaluable data; Last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 829
percentage of participants
  Baseline-Low Disease Activity | 0.36 [0.07 to 1.05]
  Week 4-Low Disease Activity | 35.98
  Week 8-Low Disease Activity | 49.57
  Week 12-Low Disease Activity | 61.75
  Week 20-Low Disease Activity | 69.25
  Week 28-Low Disease Activity | 75.79
  Week 36-Low Disease Activity | 81.96
  Baseline-Remission | 0
  Week 4-Remission | 16.52
  Week 8-Remission | 28.83
  Week 12-Remission | 38.73
  Week 20-Remission | 45.52
  Week 28-Remission | 54.24
  Week 36-Remission | 63.56

3. Secondary Outcome: Percentage of Participants Achieving DAS28 Low Disease Activity or Remission
Description: as for outcome 2
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: Period 2 (P2) mITT
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
Percentage of participants
  Week 36-Low Disease Activity | 98.5 | 99.0 | 100.0
  Week 40-Low Disease Activity | 87.8 | 84.3 | 65.4
  Week 48-Low Disease Activity | 83.1 | 81.1 | 53.3
  Week 56-Low Disease Activity | 82.6 | 81.1 | 44.7
  Week 64-Low Disease Activity | 81.6 | 82.1 | 48.7
  Week 72-Low Disease Activity | 84.1 | 82.6 | 45.7
  Week 80-Low Disease Activity | 84.6 | 81.6 | 45.7
  Week 88-Low Disease Activity | 82.6 | 80.6 | 45.2
  Week 36-Remission | 81.1 | 79.6 | 80.2
  Week 40-Remission | 68.9 | 63.5 | 42.6
  Week 48-Remission | 65.7 | 62.7 | 36.5
  Week 56-Remission | 62.2 | 65.2 | 28.9
  Week 64-Remission | 63.7 | 61.2 | 30.5
  Week 72-Remission | 67.2 | 65.2 | 27.9
  Week 80-Remission | 67.2 | 64.7 | 29.9
  Week 88-Remission | 66.7 | 60.2 | 29.4
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36 Low Disease Activity; Test type: Superiority or Other; p = 0.0853, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [0.5 to 21.4]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36 Low Disease Activity; Test type: Superiority or Other; p = 0.8491, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.2 to 4.8]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36 Low Disease Activity; Test type: Superiority or Other; p = 0.1278, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.97, 95% CI 2-sided [0.4 to 42.5]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.63, 95% CI 2-sided [2.1 to 6.4]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40 Low Disease Activity; Test type: Superiority or Other; p = 0.3027, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.8 to 2.7]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.5 to 4.2]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.55, 95% CI 2-sided [2.7 to 7.6]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48 Low Disease Activity; Test type: Superiority or Other; p = 0.5871, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.7 to 2.1]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.76, 95% CI 2-sided [2.3 to 6.1]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 6.52, 95% CI 2-sided [3.9 to 11.0]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56 Low Disease Activity; Test type: Superiority or Other; p = 0.6716, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.6 to 2.0]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.40, 95% CI 2-sided [3.4 to 8.6]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.62, 95% CI 2-sided [2.8 to 7.6]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64 Low Disease Activity; Test type: Superiority or Other; p = 0.9399, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.5 to 1.5]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.78, 95% CI 2-sided [3.0 to 7.7]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 6.25, 95% CI 2-sided [3.7 to 10.5]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72 Low Disease Activity; Test type: Superiority or Other; p = 0.6692, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.6 to 1.9]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.46, 95% CI 2-sided [3.4 to 8.7]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.74, 95% CI 2-sided [3.4 to 9.8]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80 Low Disease Activity; Test type: Superiority or Other; p = 0.4326, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.7 to 2.1]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.12, 95% CI 2-sided [3.2 to 8.2]
Statistical Analysis 22: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.68, 95% CI 2-sided [2.8 to 7.8]
Statistical Analysis 23: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88 Low Disease Activity; Test type: Superiority or Other; p = 0.6064, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.6 to 1.8]
Statistical Analysis 24: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88 Low Disease Activity; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.68, 95% CI 2-sided [3.0 to 7.4]
Statistical Analysis 25: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36 Remission; Test type: Superiority or Other; p = 0.4626, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.5 to 3.3]
Statistical Analysis 26: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36 Remission; Test type: Superiority or Other; p = 0.2886, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.6 to 3.3]
Statistical Analysis 27: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36 Remission; Test type: Superiority or Other; p = 0.7779, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.4 to 1.9]
Statistical Analysis 28: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.8 to 4.7]
Statistical Analysis 29: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40 Remission; Test type: Superiority or Other; p = 0.2091, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.8 to 2.0]
Statistical Analysis 30: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.5 to 3.6]
Statistical Analysis 31: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.33, 95% CI 2-sided [2.1 to 5.2]
Statistical Analysis 32: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48 Remission; Test type: Superiority or Other; p = 0.5351, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.7 to 1.7]
Statistical Analysis 33: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.12, 95% CI 2-sided [2.0 to 4.8]
Statistical Analysis 34: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.09, 95% CI 2-sided [2.6 to 6.5]
Statistical Analysis 35: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56 Remission; Test type: Superiority or Other; p = 0.4574, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 36: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.04, 95% CI 2-sided [3.2 to 8.0]
Statistical Analysis 37: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.19, 95% CI 2-sided [2.7 to 6.6]
Statistical Analysis 38: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64 Remission; Test type: Superiority or Other; p = 0.5229, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 39: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.84, 95% CI 2-sided [2.5 to 6.0]
Statistical Analysis 40: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.36, 95% CI 2-sided [3.3 to 8.6]
Statistical Analysis 41: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72 Remission; Test type: Superiority or Other; p = 0.6464, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 42: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.79, 95% CI 2-sided [3.0 to 7.6]
Statistical Analysis 43: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.96, 95% CI 2-sided [3.1 to 7.9]
Statistical Analysis 44: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80 Remission; Test type: Superiority or Other; p = 0.5499, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.7 to 1.7]
Statistical Analysis 45: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.11, 95% CI 2-sided [2.6 to 6.4]
Statistical Analysis 46: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.41, 95% CI 2-sided [2.8 to 7.0]
Statistical Analysis 47: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88 Remission; Test type: Superiority or Other; p = 0.1109, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.8 to 1.9]
Statistical Analysis 48: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88 Remission; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.85, 95% CI 2-sided [2.5 to 6.0]

4. Secondary Outcome: Change From Baseline in DAS28 at Weeks 4, 8, 12, 20, 28 and 36
Description: The DAS28 is a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables (the number of tender joints out of 28, the number of swollen joints out of 28 joints, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity measured on a visual analogue scale (VAS) of 100 mm). Change equals (=) Week X observation minus (-) Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; Last observation carried forward (LOCF); N=Number of participants with evaluable data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 829
units on a scale
  Baseline | 4.37 (0.02)
  Change at Week 4 | -0.88 (0.03)
  Change at Week 8 | -1.22 (0.03)
  Change at Week 12 | -1.45 (0.03)
  Change at Week 20 | -1.60 (0.03)
  Change at Week 28 | -1.72 (0.04)
  Change at Week 36 | -1.89 (0.04)

5. Secondary Outcome: Change From Week 36 in DAS28 at Weeks 40, 48, 56, 64, 72, 80 and 88
Description: The DAS28 is a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables (the number of tender joints out of 28, the number of swollen joints out of 28 joints, ESR mm/hour and PGA of disease activity measured on a VAS of 100 mm). Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; LOCF; N=number of participants with evaluable data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 196 | 197 | 188
units on a scale
  Change at Week 40 | 0.30 (0.06) | 0.31 (0.06) | 0.84 (0.06)
  Change at Week 48 | 0.40 (0.07) | 0.36 (0.07) | 1.25 (0.07)
  Change at Week 56 | 0.44 (0.07) | 0.37 (0.07) | 1.35 (0.07)
  Change at Week 64 | 0.47 (0.07) | 0.40 (0.07) | 1.33 (0.07)
  Change at Week 72 | 0.35 (0.08) | 0.38 (0.08) | 1.40 (0.08)
  Change at Week 80 | 0.40 (0.08) | 0.40 (0.08) | 1.42 (0.08)
  Change at Week 88 | 0.39 (0.08) | 0.50 (0.08) | 1.44 (0.08)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.7 to -0.4]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.9344, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.7 to -0.4]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.0 to -0.7]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.6173, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.1 to -0.7]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.1 to -0.7]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.5136, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.2 to -0.8]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.1 to -0.7]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.4868, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.1 to 0.3]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.1 to -0.7]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.3 to -0.8]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.7847, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.2 to -0.8]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.2 to -0.8]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.9810, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.2 to -0.8]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-1.3 to -0.8]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.3562, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model: Change = Week 36 score + treatment + geographic region; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.2 to -0.7]

6. Secondary Outcome: Time to Loss of Low Disease Activity DAS28 and a Change of ≥ 0.6 Units in the DAS28
Description: DAS28 calculated from the number of SJC and PJC using the 28 joints count, the ESR mm/hour and Patient's General Health VAS. VAS consisted of a line 0 to 100 mm in length; ranged from 0 (very well) to 100mm (extremely bad). Participants placed a mark indicating their health over the previous 2-3 weeks. Higher scores indicated greater affectation due to disease activity. Low disease activity = DAS28 ≤ 3.2 units. DAS28 > 3.2 to 5.1 units = moderate to high disease activity.
Time Frame: Week 36 up to Week 88
Population: P2 mITT;Imputation of failure; observed cases
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
days | NA [365.0 to NA] — NA=not applicable, median and confidence interval not estimable due to small number of occurrences of event. | NA [NA to NA] — Median and confidence interval not estimable due to small number of occurrences of event. | 85.0 [82.0 to 135.0]
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Imputation of failure defined as participants who did not reach the endpoint and discontinued due to lack of efficacy, with reason of unsatisfactory response-efficacy, adverse event, other or protocol violation were set to an event at time of discontinuation; Test type: Superiority or Other; p < 0.0001, Log Rank — Week 88 censored data was censored at 372 days
Statistical Analysis 2: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank — Week 88 censored data was censored at 372 days
Statistical Analysis 3: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.8622, Log Rank — Week 88 censored data was censored at 372 days

7. Secondary Outcome: Time to Loss of Low Disease Activity DAS28
Description: DAS28 calculated from the number of SJC and PJC using the 28 joints count, the ESR mm/hour and Patient's General Health VAS. VAS consisted of a line 0 to 100 mm in length; ranged from 0 (very well) to 100mm (extremely bad). Participants placed a mark indicating their health over the previous 2-3 weeks. Higher scores indicated greater affectation due to disease activity. DAS28 ≤ 3.2 units = low disease activity, DAS28 greater than (>)3.2 to 5.1 units = moderate to high disease activity.
Time Frame: Week 36 up to Week 88
Population: P2 mITT;
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
days | 366.0 [359.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event | NA [358.0 to NA] — Median and upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event | 85.0 [81.0 to 134.0]
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Test type: Superiority or Other; p < 0.0001, Log Rank — Week 88 censored data was censored at 372 days
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Test type: Superiority or Other; p = 0.9841, Log Rank — Week 88 censored data was censored at 372 days
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Test type: Superiority or Other; p < 0.0001, Log Rank — Week 88 censored data was censored at 372 days

8. Secondary Outcome: Proportion of Time Participants Had Low Disease Activity DAS28 Week 36 to Week 88
Description: DAS28 calculated from the number of SJC and PJC using the 28 joints, the ESR mm/hour and Patient's General Health VAS. VAS consisted of a line 0 to 100 mm in length; ranged from 0 (very well) to 100mm (extremely bad). Participants placed a mark indicating their health over the previous 2-3 weeks. Higher scores indicated greater affectation due to disease activity. DAS28 < 3.2 units = low disease activity. Cumulative proportion calculated as time-averaged Area Under the Curve (AUC) (AUC divided by number of weeks at that time point), with AUC calculated from Week 36 and Week 88.
Time Frame: Week 36 up to Week 88
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: proportion of weeks in DAS28 <3.2
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
proportion of weeks in DAS28 <3.2 | 0.85 (0.02) | 0.84 (0.02) | 0.58 (0.02)

9. Secondary Outcome: Change From Baseline in Prorated Swollen Joint Count at Weeks 4, 8, 12, 20, 28 and 36
Description: American College of Rheumatology (ACR), swollen joint count were an assessment of 28 joints. Joints are classified as either swollen or not swollen. If < 20% of swollen joints missing then total swollen joint prorated (multiplied by 28 divided by (/) number of non-missing swollen joints). Total possible score ranged from -28 to 28. An increase in swollen joints from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression and a decrease represented improvement. Change = Week X observation - baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Error); unit: number of swollen joints
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 830
number of swollen joints
  Baseline | 3.82 (0.09)
  Change at Week 4 | -1.31 (0.08)
  Change at Week 8 | -1.96 (0.08)
  Change at Week 12 | -2.29 (0.08)
  Change at Week 20 | -2.60 (0.09)
  Change at Week 28 | -2.70 (0.09)
  Change at Week 36 | -2.67 (0.10)

10. Secondary Outcome: Prorated Swollen Joint Count at Week 36
Description: ACR, swollen joint count was an assessment of 28 joints. Joints were classified as either swollen or not swollen. If < 20% of swollen joints missing then total swollen joint prorated (multiplied by 28 divided by number of non-missing swollen joints). Total possible score of swollen joints ranged from 0-28.
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: number of swollen joints
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
number of swollen joints | 0.63 (0.11) | 0.57 (0.09) | 0.59 (0.08)

11. Secondary Outcome: Change From Week 36 in Prorated Swollen Joint Count at Weeks 40, 48, 56, 64, 72, 80 and 88
Description: ACR, swollen joint count was an assessment of 28 joints. Joints were classified as either swollen or not swollen. If < 20% of swollen joints missing then total swollen joint prorated (multiplied by 28 divided by (/) number of non-missing swollen joints). Total possible score ranged from -28 to 28. An increase in swollen joints from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression and a decrease represented improvement. Change = Week X observation - Week 36 observation.
Time Frame: Week 36, Weeks 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: number of swollen joints
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
number of swollen joints
  Change at Week 40 | 0.10 (0.11) | 0.14 (0.11) | 0.91 (0.11)
  Change at Week 48 | 0.25 (0.15) | 0.21 (0.15) | 1.38 (0.15)
  Change at Week 56 | 0.28 (0.16) | 0.26 (0.16) | 1.49 (0.16)
  Change at Week 64 | 0.37 (0.17) | 0.34 (0.17) | 1.64 (0.17)
  Change at Week 72 | 0.20 (0.16) | 0.22 (0.16) | 1.64 (0.17)
  Change at Week 80 | 0.25 (0.18) | 0.32 (0.18) | 1.82 (0.18)
  Change at Week 88 | 0.17 (0.18) | 0.49 (0.18) | 1.92 (0.18)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model: Change = Week 36 score + treatment + geographic region + DAS28 Strata. DAS28 Strata is defined as DAS28 low disease (≤3.2) or remission (<2.6) at randomization; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.8015, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-1.5 to -0.7]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.8534, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-1.6 to -0.8]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-1.7 to -0.8]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.9074, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-1.7 to -0.8]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-1.8 to -0.8]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.9229, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-1.8 to -0.8]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-1.9 to -1.0]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.9279, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-1.9 to -1.0]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-2.1 to -1.1]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.7695, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.6 to 0.4]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-2.0 to -1.0]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-2.3 to -1.2]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.2182, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.8 to 0.2]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-1.9 to -0.9]

12. Secondary Outcome: Change From Baseline in the Painful Joint Count at Weeks 4, 8, 12, 20, 28 and 36
Description: A total of 28 joints were assessed by the investigator using criteria based on pressure and joint manipulation. Total possible scores ranged from -28 to 28. An increase in joint pain count from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression and a decrease represented improvement. Change = Week X observation - Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Error); unit: number of painful joints
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 830
number of painful joints
  Baseline | 5.09 (0.10)
  Change at Week 4 | -1.68 (0.10)
  Change at Week 8 | -2.50 (0.10)
  Change at Week 12 | -2.86 (0.11)
  Change at Week 20 | -3.11 (0.12)
  Change at Week 28 | -3.32 (0.12)
  Change at Week 36 | -3.51 (0.13)

13. Secondary Outcome: Painful Joint Count at Week 36
Description: A total of 28 joints were assessed by the investigator using criteria based on pressure and joint manipulation. Total possible score ranged form 0-28.
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: number of painful joints
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
number of painful joints | 0.64 (0.08) | 0.69 (0.09) | 0.74 (0.09)

14. Secondary Outcome: Change From Week 36 in Painful Joint Count at Weeks 40, 48, 56, 64, 72, 80 and 88
Description: Total of 28 joints were assessed by the investigator using criteria based on pressure and joint manipulation. Total possible scores ranged from -28 to 28. An increase in joint pain count from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression and a decrease represented improvement. Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Least Squares Mean (Standard Error); unit: number of painful joints
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 196 | 197 | 188
number of painful joints
  Change at Week 40 | 0.61 (0.17) | 0.49 (0.17) | 1.47 (0.17)
  Change at Week 48 | 0.67 (0.21) | 0.63 (0.21) | 2.69 (0.21)
  Change at Week 56 | 0.61 (0.20) | 0.66 (0.20) | 2.67 (0.21)
  Change at Week 64 | 0.79 (0.22) | 0.73 (0.22) | 2.76 (0.22)
  Change at Week 72 | 0.63 (0.23) | 0.78 (0.23) | 3.01 (0.23)
  Change at Week 80 | 0.74 (0.23) | 0.88 (0.23) | 3.02 (0.23)
  Change at Week 88 | 0.73 (0.24) | 0.78 (0.24) | 3.14 (0.24)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.3 to -0.4]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.6088, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.4 to -0.5]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.02, 95% CI 2-sided [-2.6 to -1.4]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.9048, ANOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-2.6 to -1.5]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-2.6 to -1.5]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.8437, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-2.6 to -1.4]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.6 to -1.4]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.8587, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.6 to 0.7]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-2.6 to -1.4]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.38, 95% CI 2-sided [-3.0 to -1.8]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.6323, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.23, 95% CI 2-sided [-2.9 to -1.6]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-2.9 to -1.6]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.6558, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-2.8 to -1.5]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-3.1 to -1.7]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.8688, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-3.0 to -1.7]

15. Secondary Outcome: Change From Baseline in the Physician Global Assessment (PGA) at Weeks 4, 8, 12, 20, 28 and 36
Description: PGA of Disease Activity was measured on a 0 to 10 Scale, with 0 = no disease activity and 10 = extreme disease activity. Change = Week X observation - Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 833
units on a scale
  Baseline | 4.11 (0.05)
  Change at Week 4 | -1.29 (0.05)
  Change at Week 8 | -1.84 (0.06)
  Change at Week 12 | -2.09 (0.06)
  Change at Week 20 | -2.26 (0.06)
  Change at Week 28 | -2.45 (0.06)
  Change at Week 36 | -2.57 (0.06)

16. Secondary Outcome: PGA Score at Week 36
Description: PGA of Disease Activity was measured on a 0 to 10 Scale, with 0 = no disease activity and 10 = extreme disease activity.
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
units on a scale | 1.06 (0.07) | 1.19 (0.08) | 1.11 (0.05)

17. Secondary Outcome: Change From Week 36 in the PGA Score at Weeks 40, 48, 56, 64, 72, 80 and 88
Description: PGA of Disease Activity was measured on a 0 to 10 Scale, with 0 = no disease activity and 10 = extreme disease activity. Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
units on a scale
  Change at Week 40 | 0.25 (0.09) | 0.24 (0.09) | 0.98 (0.09)
  Change at Week 48 | 0.37 (0.10) | 0.26 (0.11) | 1.48 (0.11)
  Change at Week 56 | 0.37 (0.10) | 0.34 (0.10) | 1.49 (0.11)
  Change at Week 64 | 0.41 (0.11) | 0.26 (0.11) | 1.51 (0.11)
  Change at Week 72 | 0.32 (0.11) | 0.24 (0.11) | 1.57 (0.11)
  Change at Week 80 | 0.27 (0.11) | 0.34 (0.11) | 1.61 (0.11)
  Change at Week 88 | 0.23 (0.11) | 0.35 (0.12) | 1.67 (0.12)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.0 to -0.5]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.9636, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.0 to -0.5]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-1.4 to -0.8]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.4605, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-1.5 to -0.9]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-1.4 to -0.8]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.8404, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.4 to -0.9]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.4 to -0.8]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.3118, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-1.6 to -1.0]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-1.6 to -0.9]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.6100, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.2 to 0.4]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-1.6 to -1.0]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-1.6 to -1.0]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.6552, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-1.6 to -1.0]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-1.8 to -1.1]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.4753, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-1.6 to -1.0]

18. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PtGA) of Arthritis Pain at Weeks 4, 8, 12, 20, 28 and 36
Description: Participants asked to rate their overall arthritis activity by circling a number ranging from 0 (no disease activity) to 10 (extreme disease activity). Change = Week X observation - Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 832
units on a scale
  Baseline | 4.85 (0.06)
  Change at Week 4 | -1.16 (0.06)
  Change at Week 8 | -1.46 (0.07)
  Change at Week 12 | -1.68 (0.07)
  Change at Week 20 | -2.01 (0.07)
  Change at Week 28 | -2.14 (0.08)
  Change at Week 36 | -2.46 (0.08)

19. Secondary Outcome: PtGA of Arthritis Pain at Week 36
Description: PtGA asked the participant to assess their overall arthritis activity. Participants responded by circling a number ranging from 0 (no disease activity) to 10 (extreme disease activity).
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
units on a scale | 1.80 (0.12) | 1.77 (0.10) | 1.86 (0.11)

20. Secondary Outcome: Change From Week 36 in PtGA of Arthritis Pain at Weeks 40, 48, 56, 64, 72, 80, 88
Description: PtGA asked the participant to assess their overall arthritis activity. Participants responded by circling a number ranging from 0 (no disease activity) to 10 (extreme disease activity). Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80, 88
Population: P2 mITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
units on a scale
  Change at Week 40 | 0.41 (0.12) | 0.46 (0.11) | 1.28 (0.12)
  Change at Week 48 | 0.36 (0.12) | 0.54 (0.12) | 1.76 (0.13)
  Change at Week 56 | 0.47 (0.13) | 0.60 (0.13) | 1.76 (0.13)
  Change at Week 64 | 0.45 (0.13) | 0.60 (0.13) | 1.75 (0.13)
  Change at Week 72 | 0.33 (0.14) | 0.67 (0.14) | 1.93 (0.14)
  Change at Week 80 | 0.15 (0.13) | 0.57 (0.13) | 1.70 (0.13)
  Change at Week 88 | 0.29 (0.14) | 0.59 (0.14) | 1.84 (0.14)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.2 to -0.6]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.7427, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.40, 95% CI 2-sided [-1.7 to -1.1]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.3129, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.6 to -0.9]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.6 to -0.9]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.4645, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-1.5 to -0.8]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.30, 95% CI 2-sided [-1.7 to -0.9]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.3793, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.5 to 0.2]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-1.5 to -0.8]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-2.0 to -1.2]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.0816, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.7 to 0.0]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-1.6 to -0.9]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-1.9 to -1.2]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.0256, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.8 to -0.1]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-1.5 to -0.8]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-1.9 to -1.2]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.1158, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.7 to 0.1]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-1.6 to -0.9]

21. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Weeks 4, 8, 12, 20, 28 and 36
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and when the participants were able to resume normal activities without stiffness. No stiffness present = 0; stiffness persisted the entire day = 1440 minutes (24 hour times [*] 60 min) was recorded. Change = Week X observation - Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Deviation); unit: minutes (min)
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 830
minutes (min)
  Baseline | 176.98 (333.51)
  Change at Week 4 | -81.31 (335.75)
  Change at Week 8 | -80.73 (342.65)
  Change at Week 12 | -90.64 (380.18)
  Change at Week 20 | -101.75 (378.01)
  Change at Week 28 | -97.85 (377.65)
  Change at Week 36 | -112.36 (358.94)

22. Secondary Outcome: Duration of Morning Stiffness at Week 36
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and when the participants were able to resume normal activities without stiffness. No stiffness present = 0; stiffness persisted the entire day = 1440 minutes (24 hour * 60 min) was recorded.
Time Frame: Week 36
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Error); unit: min
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 200 | 201 | 196
min | 34.60 (10.35) | 36.46 (8.13) | 38.03 (10.84)

23. Secondary Outcome: Change From Week 36 in Duration of Morning Stiffness at Weeks 40, 48, 56, 64, 72, 80, 88
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness. No stiffness present = 0; stiffness persisted the entire day = 1440 minutes (24 hour * 60 min) was recorded. Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80, 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Least Squares Mean (Standard Error); unit: min
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 200 | 201 | 196
min
  Change at Week 40 | 3.43 (12.82) | 14.00 (12.60) | 45.10 (12.83)
  Change at Week 48 | -7.64 (14.47) | 35.54 (14.47) | 72.41 (14.62)
  Change at Week 56 | -2.10 (14.19) | 24.04 (14.19) | 87.09 (14.34)
  Change at Week 64 | 13.80 (16.09) | 15.65 (16.10) | 98.16 (16.26)
  Change at Week 72 | 8.30 (17.36) | 18.50 (17.37) | 117.04 (17.54)
  Change at Week 80 | -1.06 (15.18) | 12.63 (15.18) | 114.42 (15.34)
  Change at Week 88 | 24.54 (16.29) | 12.23 (16.30) | 96.14 (16.46)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0214, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -41.67, 95% CI 2-sided [-77.1 to -6.2]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.5544, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -10.57, 95% CI 2-sided [-45.6 to 24.5]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0826, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -31.10, 95% CI 2-sided [-66.2 to 4.0]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -80.05, 95% CI 2-sided [-120.3 to -39.8]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.0344, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -43.18, 95% CI 2-sided [-83.2 to -3.2]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.0721, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -36.87, 95% CI 2-sided [-77.1 to 3.3]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -89.19, 95% CI 2-sided [-128.7 to -49.7]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.1910, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -26.14, 95% CI 2-sided [-65.4 to 13.1]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.0018, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -63.05, 95% CI 2-sided [-102.5 to -23.6]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -84.36, 95% CI 2-sided [-129.1 to -39.6]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.9350, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-46.3 to 42.6]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -82.52, 95% CI 2-sided [-127.2 to -37.8]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -108.73, 95% CI 2-sided [-157.0 to -60.4]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.6764, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -10.20, 95% CI 2-sided [-58.2 to 37.8]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -98.53, 95% CI 2-sided [-146.7 to -50.3]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -115.48, 95% CI 2-sided [-157.7 to -73.3]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.5219, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -13.69, 95% CI 2-sided [-55.6 to 28.3]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -101.80, 95% CI 2-sided [-144.0 to -59.6]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.0020, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -71.60, 95% CI 2-sided [-116.9 to -26.3]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.5917, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = 12.30, 95% CI 2-sided [-32.7 to 57.3]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -83.91, 95% CI 2-sided [-129.2 to -38.7]

24. Secondary Outcome: Change From Baseline in General Health at Weeks 4, 8, 12, 20, 28 and 36
Description: General Health VAS is a 100 millimeter (mm) line marked by the participant. Participants were asked, "In general how would you rate your health over the last 2 to 3 weeks?" Scores ranged from 0 mm = very well to 100 mm = extremely bad. Change = Week X observation - Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 832
mm
  Baseline | 43.37 (16.95)
  Change at Week 4 | -9.39 (18.93)
  Change at Week 8 | -12.36 (21.17)
  Change at Week 12 | -15.69 (20.72)
  Change at Week 20 | -18.65 (21.09)
  Change at Week 28 | -19.47 (22.47)
  Change at Week 36 | -22.66 (22.06)

25. Secondary Outcome: General Health at Week 36
Description: General Health VAS is a 100 mm line marked by the participant. Participants are asked, "In general how would you rate your health over the last 2 to 3 weeks?" Scores ranged from 0 mm = very well to 100 mm = extremely bad.
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
mm | 14.12 (1.11) | 14.77 (1.06) | 15.09 (1.10)

26. Secondary Outcome: Change From Week 36 in General Health at Weeks 40, 48, 56, 64, 72, 80, 88
Description: General Health VAS is a 100 mm line marked by the participant. Participants were asked, "In general how would you rate your health over the last 2 to 3 weeks?" Scores ranged from 0 mm = very well to 100 mm = extremely bad. Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80, 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 196
mm
  Change at Week 40 | 3.26 (1.12) | 5.82 (1.11) | 12.05 (1.13)
  Change at Week 48 | 4.67 (1.19) | 5.36 (1.20) | 16.76 (1.21)
  Change at Week 56 | 5.09 (1.25) | 6.46 (1.26) | 17.19 (1.27)
  Change at Week 64 | 4.04 (1.22) | 5.36 (1.22) | 16.87 (1.23)
  Change at Week 72 | 3.76 (1.33) | 6.88 (1.33) | 18.55 (1.34)
  Change at Week 80 | 2.70 (1.28) | 4.59 (1.28) | 17.26 (1.29)
  Change at Week 88 | 3.89 (1.33) | 6.22 (1.33) | 17.06 (1.34)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -8.79, 95% CI 2-sided [-11.9 to -5.7]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.1033, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-5.6 to 0.5]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -6.23, 95% CI 2-sided [-9.3 to -3.1]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.09, 95% CI 2-sided [-15.4 to -8.8]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.6802, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-4.0 to 2.6]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -11.39, 95% CI 2-sided [-14.7 to -8.1]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.09, 95% CI 2-sided [-15.6 to -8.6]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.4404, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-4.8 to 2.1]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -10.73, 95% CI 2-sided [-14.2 to -7.2]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.83, 95% CI 2-sided [-16.2 to -9.4]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.4437, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-4.7 to 2.1]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -11.51, 95% CI 2-sided [-14.9 to -8.1]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -14.79, 95% CI 2-sided [-18.5 to -11.1]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.0960, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-6.8 to 0.6]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -11.67, 95% CI 2-sided [-15.4 to -8.0]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -14.56, 95% CI 2-sided [-18.1 to -11.0]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.2948, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-5.4 to 1.6]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.68, 95% CI 2-sided [-16.2 to -9.1]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -13.16, 95% CI 2-sided [-16.9 to -9.5]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.2130, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.33, 95% CI 2-sided [-6.0 to 1.3]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -10.83, 95% CI 2-sided [-14.5 to -7.1]

27. Secondary Outcome: Change From Baseline in Pain at Weeks 4, 8, 12, 20, 28 and 36
Description: 100 mm line (Visual Analog Scale) marked by participant. Intensity of pain range (over past 2 to 3 days): 0 = no pain to 100 = worst possible pain. Change = Week X observation - Baseline observation.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 832
mm
  Baseline | 45.47 (0.60)
  Change at Week 4 | -13.06 (0.69)
  Change at Week 8 | -17.11 (0.73)
  Change at Week 12 | -19.47 (0.73)
  Change at Week 20 | -22.11 (0.73)
  Change at Week 28 | -22.98 (0.78)
  Change at Week 36 | -25.96 (0.76)

28. Secondary Outcome: Pain at Week 36
Description: 100 mm line (Visual Analog Scale) marked by participant. Intensity of pain range (over past 2 to 3 days): 0 = no pain to 100 = pain as bad as it could be. Change = Week x observation minus (-) Baseline observation.
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
mm | 12.78 (1.09) | 13.87 (1.04) | 14.21 (1.11)

29. Secondary Outcome: Change From Week 36 in Pain at Weeks 40, 48, 56, 64, 72, 80 and 88
Description: 100 mm line (Visual Analog Scale) marked by participant. Intensity of pain range (over past 2 to 3 days): 0 = no pain to 100 = worst possible pain. Change = Week X observation - Week 36 observation.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
mm
  Change at Week 40 | 4.50 (1.15) | 4.91 (1.15) | 13.05 (1.17)
  Change at Week 48 | 5.16 (1.29) | 5.66 (1.30) | 18.77 (1.31)
  Change at Week 56 | 5.23 (1.29) | 6.25 (1.29) | 17.76 (1.30)
  Change at Week 64 | 4.61 (1.32) | 6.55 (1.32) | 18.49 (1.33)
  Change at Week 72 | 4.26 (1.37) | 7.05 (1.37) | 19.90 (1.38)
  Change at Week 80 | 3.36 (1.36) | 5.92 (1.36) | 18.23 (1.37)
  Change at Week 88 | 3.88 (1.37) | 6.31 (1.37) | 18.57 (1.39)
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -8.55, 95% CI 2-sided [-11.8 to -5.3]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.8033, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-3.6 to 2.8]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -8.14, 95% CI 2-sided [-11.3 to -4.9]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -13.61, 95% CI 2-sided [-17.2 to -10.0]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.7830, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-4.1 to 3.1]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -13.11, 95% CI 2-sided [-16.7 to -9.5]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.53, 95% CI 2-sided [-16.1 to -8.9]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.5732, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-4.6 to 2.5]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -11.50, 95% CI 2-sided [-15.1 to -7.9]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -13.88, 95% CI 2-sided [-17.6 to -10.2]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.2972, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -1.94, 95% CI 2-sided [-5.6 to 1.7]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -11.94, 95% CI 2-sided [-15.6 to -8.3]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -15.64, 95% CI 2-sided [-19.4 to -11.8]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.1477, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.80, 95% CI 2-sided [-6.6 to 1.0]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.85, 95% CI 2-sided [-16.6 to -9.0]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -14.87, 95% CI 2-sided [-18.6 to -11.1]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.1808, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-6.3 to 1.2]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.31, 95% CI 2-sided [-16.1 to -8.5]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -14.70, 95% CI 2-sided [-18.5 to -10.9]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.2077, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -2.44, 95% CI 2-sided [-6.2 to 1.4]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Final Values) = -12.26, 95% CI 2-sided [-16.1 to -8.5]

30. Secondary Outcome: Percentage of Participants Achieving an Acceptable State on the Patient Acceptable Symptom State (PASS) at Baseline and Week 36
Description: PASS was a 1 question assessment of how rheumatoid arthritis has affected the participant in the last 2 days (If you were to remain in the next few months as you were during the last 2 days, would this be acceptable or unacceptable to you?).
Time Frame: Baseline, Week 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 824
percentage of participants
  Baseline | 44.90 [41.47 to 48.37]
  Week 36 | 86.80 [84.26 to 89.06]
Statistical Analysis 1: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel

31. Secondary Outcome: Percentage of Participants Achieving an Acceptable State on the PASS at Week 36 and Weeks 64 and 88
Description: as for outcome 30
Time Frame: Weeks 36, 64 and 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 188 | 178 | 185
percentage of participants
  Week 36 | 93.5 | 89.9 | 93.9
  Week 64 | 90.0 | 88.7 | 65.8
  Week 88 | 91.3 | 84.7 | 70.1
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.8974, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.5 to 2.5]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.1105, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.8 to 3.7]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.1900, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.3 to 1.4]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.18, 95% CI 2-sided [2.3 to 7.5]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.4032, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.6 to 2.4]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.23, 95% CI 2-sided [2.4 to 7.5]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [2.1 to 7.2]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.0272, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.0 to 3.6]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.4 to 4.0]

32. Secondary Outcome: Percentage of Participants Achieving European League Against Rheumatism (EULAR) Good or Moderate Response at Weeks 4, 8, 12, 20, 28 and 36
Description: EULAR Response Criteria: Good response was defined as >1.2 units improvement in DAS28 from Baseline and DAS28 attained up to Week 88 of <=3.2 units. Non responders were participants with improvement of <0.6 units or participants with improvement of 0.6 to 1.2 units and DAS28 attained up to Week 88 of > 5.1 units. Remaining participants were defined as having a moderate response. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 823
percentage of participants
  Week 4 | 61.95 [58.44 to 65.38]
  Week 8 | 75.37
  Week 12 | 82.03
  Week 20 | 86.63
  Week 28 | 87.24
  Week 36 | 87.97
Statistical Analysis 1: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 28; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 36; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

33. Secondary Outcome: Percentage of Participants Achieving EULAR Good or Moderate Response at Week 36, 40, 48, 56, 64, 72, 80 and 88
Description: as for outcome 32
Time Frame: Week 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 198 | 199 | 191
percentage of participants
  Week 36 | 99.0 | 99.0 | 97.5
  Week 40 | 93.8 | 95.4 | 76.1
  Week 48 | 91.0 | 92.0 | 64.0
  Week 56 | 90.0 | 91.5 | 64.5
  Week 64 | 92.0 | 91.5 | 62.4
  Week 72 | 93.0 | 89.1 | 61.4
  Week 80 | 92.0 | 89.1 | 60.4
  Week 88 | 90.5 | 88.1 | 61.9
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.1718, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.5 to 10.7]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.8303, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.2 to 7.3]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.2130, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.27, 95% CI 2-sided [0.5 to 10.1]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.10, 95% CI 2-sided [2.1 to 8.2]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.4337, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.3 to 2.0]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.14, 95% CI 2-sided [2.5 to 10.8]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.61, 95% CI 2-sided [3.0 to 10.5]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.8973, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.4 to 1.9]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.33, 95% CI 2-sided [2.8 to 10.1]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.4 to 8.1]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.5708, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.4 to 1.7]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.58, 95% CI 2-sided [3.0 to 10.3]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 6.29, 95% CI 2-sided [3.3 to 12.0]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.8842, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.4 to 2.0]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 5.92, 95% CI 2-sided [3.2 to 10.8]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 7.39, 95% CI 2-sided [3.8 to 14.4]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.1608, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.6 to 3.1]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.92, 95% CI 2-sided [2.9 to 8.4]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 6.44, 95% CI 2-sided [3.4 to 12.4]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.2825, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.6 to 2.7]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.59, 95% CI 2-sided [2.7 to 7.8]
Statistical Analysis 22: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.81, 95% CI 2-sided [2.7 to 8.7]
Statistical Analysis 23: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.4471, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.5 to 2.1]
Statistical Analysis 24: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.19, 95% CI 2-sided [2.5 to 7.0]

34. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20 Percent (%) (ACR20) Response at Weeks 4, 8, 12, 20, 28 and 36
Description: ACR20 response, ≥ 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and = at least 20% improvement in at least 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant (ESR).
Time Frame: Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 824
percentage of participants
  Week 4 | 38.62
  Week 8 | 53.14
  Week 12 | 61.29
  Week 20 | 66.87
  Week 28 | 70.75
  Week 36 | 72.82
Statistical Analysis 1: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 28; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 36; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

35. Secondary Outcome: Percentage of Participants With an ACR20 Response at Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Description: ACR20 response: ≥ 20% improvement in tender joint count; ≥20% improvement in swollen joint count; and = at least 20% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; LOCF; N=number of participants with evaluable data
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 200 | 201 | 197
percentage of participants
  Week 36 | 86.5 | 85.1 | 88.3
  Week 40 | 76.9 | 77.7 | 61.2
  Week 48 | 77.0 | 76.1 | 50.3
  Week 56 | 75.0 | 74.6 | 50.3
  Week 64 | 76.5 | 74.1 | 48.7
  Week 72 | 78.0 | 74.6 | 47.2
  Week 80 | 79.5 | 77.6 | 46.7
  Week 88 | 75.5 | 74.6 | 48.7
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.6006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.4 to 1.6]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.4967, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.6 to 2.1]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.3648, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.4 to 1.5]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0024, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.2 to 3.2]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.8308, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.92, 95% CI [0.6 to 1.]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.3 to 3.4]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.25, 95% CI 2-sided [2.0 to 5.2]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.7374, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.9 to 4.8]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.9 to 4.8]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.9599, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.9 to 4.6]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.59, 95% CI 2-sided [2.3 to 5.7]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.4509, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.8 to 2.0]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.9 to 4.6]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.28, 95% CI 2-sided [2.6 to 7.0]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.3037, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.7 to 2.0]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.27, 95% CI 2-sided [2.1 to 5.1]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.41, 95% CI 2-sided [2.7 to 7.2]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.6076, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.7 to 1.9]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.80, 95% CI 2-sided [2.4 to 6.0]
Statistical Analysis 22: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.85, 95% CI 2-sided [1.8 to 4.6]
Statistical Analysis 23: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.7837, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.6 to 1.6]
Statistical Analysis 24: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [2.0 to 4.7]

36. Secondary Outcome: Percentage of Participants With an ACR50 Response at Weeks 4, 8, 12, 20, 28 and 36
Description: ACR50 response: ≥ 50% improvement in tender joint count; = ≥50% improvement in swollen joint count; and = at least 50% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).
Time Frame: Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 824
percentage of participants
  Week 4 | 11.25
  Week 8 | 22.88
  Week 12 | 31.99
  Week 20 | 41.99
  Week 28 | 51.33
  Week 36 | 59.83
Statistical Analysis 1: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 28; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 36; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

37. Secondary Outcome: Percentage of Participants With an ACR50 Response at Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Description: as for outcome 36
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 200 | 201 | 197
percentage of participants
  Week 36 | 76.5 | 70.6 | 74.1
  Week 40 | 60.5 | 57.9 | 41.0
  Week 48 | 58.0 | 59.2 | 33.5
  Week 56 | 62.0 | 56.2 | 28.9
  Week 64 | 59.0 | 55.7 | 27.9
  Week 72 | 63.0 | 53.7 | 26.9
  Week 80 | 62.5 | 58.7 | 27.4
  Week 88 | 62.5 | 57.2 | 25.9
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.5263, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.7 to 2.0]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.1055, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.9 to 2.3]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.4348, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.4 to 3.3]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.5511, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.7 to 1.7]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.3 to 2.9]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.79, 95% CI 2-sided [1.8 to 4.3]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.9225, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.6 to 1.5]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.95, 95% CI 2-sided [1.9 to 4.5]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.20, 95% CI 2-sided [2.7 to 6.6]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.2454, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.9 to 2.0]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.15, 95% CI 2-sided [2.0 to 4.9]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.83, 95% CI 2-sided [2.4 to 6.0]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.4919, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.8 to 1.9]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.16, 95% CI 2-sided [2.0 to 4.9]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.80, 95% CI 2-sided [3.0 to 7.6]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.0658, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.0 to 2.3]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [2.0 to 4.7]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.32, 95% CI 2-sided [2.7 to 6.8]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.4014, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.8 to 1.9]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.54, 95% CI 2-sided [2.3 to 5.5]
Statistical Analysis 22: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.53, 95% CI 2-sided [2.9 to 7.2]
Statistical Analysis 23: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.2824, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.8 to 1.9]
Statistical Analysis 24: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.83, 95% CI 2-sided [2.5 to 5.9]

38. Secondary Outcome: Percentage of Participants With an ACR70 Response at Weeks 4, 8, 12, 20, 28 and 36
Description: ACR70 response: ≥ 70% improvement in tender joint count; = ≥70% improvement in swollen joint count; and = at least 70% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).
Time Frame: Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 824
percentage of participants
  Week 4 | 2.81
  Week 8 | 6.77
  Week 12 | 10.26
  Week 20 | 16.75
  Week 28 | 22.45
  Week 36 | 27.79
Statistical Analysis 1: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 28; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; week 36; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

39. Secondary Outcome: Percentage of Participants With an ACR70 Response at Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Description: ACR70 response: ≥ 70% improvement in tender joint count; = ≥70% improvement in swollen joint count; and = at least 70% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and C-Reactive Protein CRP.
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; N=number of participants with evaluable data; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 200 | 201 | 197
percentage of participants
  Week 36 | 42.0 | 33.3 | 33.0
  Week 40 | 28.7 | 27.9 | 17.6
  Week 48 | 28.0 | 30.8 | 9.6
  Week 56 | 31.0 | 31.3 | 10.2
  Week 64 | 33.0 | 28.9 | 10.2
  Week 72 | 32.0 | 31.3 | 10.7
  Week 80 | 34.0 | 30.3 | 10.7
  Week 88 | 35.5 | 31.3 | 11.2
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.0575, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.0 to 2.3]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.0630, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.0 to 2.3]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.9160, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.7 to 1.6]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0147, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.0 to 3.0]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.8675, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.6 to 1.6]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0174, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.1 to 3.0]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.9 to 5.7]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.4941, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 4.01, 95% CI 2-sided [2.3 to 7.0]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.40, 95% CI 2-sided [2.0 to 5.9]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.8185, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.6 to 1.5]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [2.1 to 6.4]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.78, 95% CI 2-sided [2.2 to 6.6]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.4254, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.38, 95% CI 2-sided [1.9 to 5.9]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.8 to 5.8]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.8766, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.7 to 1.6]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [2.1 to 6.4]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.53, 95% CI 2-sided [2.0 to 6.4]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.3535, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.8 to 1.9]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.44, 95% CI 2-sided [1.9 to 6.1]
Statistical Analysis 22: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.45, 95% CI 2-sided [2.0 to 6.1]
Statistical Analysis 23: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.3231, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.8 to 1.9]
Statistical Analysis 24: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.23, 95% CI 2-sided [1.9 to 5.6]

40. Secondary Outcome: Percentage of Participants With an ACR90 Response at Weeks 4, 8, 12, 20, 28 and 36
Description: ACR90 response: ≥ 90% improvement in tender joint count; = ≥90% improvement in swollen joint count; and = at least 90% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).
Time Frame: Weeks 4, 8, 12, 20, 28 and 36
Population: P1 mITT; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1
Number analyzed (Participants) | 824
percentage of participants
  Week 4 | 1.02
  Week 8 | 1.23
  Week 12 | 1.83
  Week 20 | 4.13
  Week 28 | 6.31
  Week 36 | 8.25
Statistical Analysis 1: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 28; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1; Week 36; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

41. Secondary Outcome: Percentage of Participants With an ACR90 Response at Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Description: ACR90 response: ≥ 90% improvement in tender joint count; = 90% improvement in swollen joint count; and = 90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).
Time Frame: Weeks 36, 40, 48, 56, 64, 72, 80 and 88
Population: P2 mITT; LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 200 | 201 | 197
percentage of participants
  Week 36 | 13.5 | 14.4 | 5.6
  Week 40 | 10.3 | 9.1 | 4.8
  Week 48 | 10.0 | 9.5 | 2.5
  Week 56 | 9.5 | 9.0 | 2.0
  Week 64 | 10.5 | 11.9 | 2.5
  Week 72 | 12.0 | 13.9 | 2.5
  Week 80 | 14.0 | 12.9 | 3.0
  Week 88 | 17.0 | 14.4 | 3.6
Statistical Analysis 1: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.0089, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.14, 95% CI 2-sided [0.9 to 5.2]
Statistical Analysis 2: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.6932, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.5 to 1.7]
Statistical Analysis 3: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 36; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.2 to 6.1]
Statistical Analysis 4: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0797, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.6 to 3.6]
Statistical Analysis 5: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.8103, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.4 to 1.9]
Statistical Analysis 6: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 40; Test type: Superiority or Other; p = 0.0903, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.8 to 4.5]
Statistical Analysis 7: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.2 to 7.8]
Statistical Analysis 8: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.9770, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.5 to 2.0]
Statistical Analysis 9: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 48; Test type: Superiority or Other; p = 0.0036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.3 to 8.3]
Statistical Analysis 10: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.0038, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.0 to 7.7]
Statistical Analysis 11: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.9055, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.5 to 2.0]
Statistical Analysis 12: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 56; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.2 to 9.8]
Statistical Analysis 13: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.35, 95% CI 2-sided [1.3 to 8.8]
Statistical Analysis 14: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.5763, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.4 to 1.7]
Statistical Analysis 15: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 64; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.93, 95% CI 2-sided [1.5 to 10.0]
Statistical Analysis 16: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.21, 95% CI 2-sided [1.2 to 8.8]
Statistical Analysis 17: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p = 0.4828, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.4 to 1.6]
Statistical Analysis 18: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 72; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.52, 95% CI 2-sided [1.4 to 9.0]
Statistical Analysis 19: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.4 to 7.8]
Statistical Analysis 20: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.8553, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.6 to 1.9]
Statistical Analysis 21: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 80; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.56, 95% CI 2-sided [1.5 to 8.7]
Statistical Analysis 22: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.53, 95% CI 2-sided [1.6 to 7.6]
Statistical Analysis 23: Comparison: Etanercept 50 mg Plus MTX -Period 2 vs Etanercept 25 mg Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.5025, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.6 to 2.0]
Statistical Analysis 24: Comparison: Etanercept 25 mg Plus MTX-Period 2 vs Placebo Plus MTX-Period 2; Week 88; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 3.62, 95% CI 2-sided [1.6 to 8.1]

42. Secondary Outcome: DAS28 at Week 36
Description: The DAS28 is a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables (the number of tender joints out of 28, the number of swollen joints out of 28 joints, ESR mm/hour and PGA of disease activity measured on a VAS of 100 mm).
Time Frame: Week 36
Population: P2 mITT; LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Number analyzed (Participants) | 201 | 201 | 197
units on a scale | 1.99 (0.04) | 2.06 (0.04) | 2.07 (0.04)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participants and as nonserious in another participants, or one participants may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1 | Etanercept 50 mg Plus MTX -Period 2 | Etanercept 25 mg Plus MTX-Period 2 | Placebo Plus MTX-Period 2
Serious Adverse Events (participants affected / at risk) | 38/834 | 13/202 | 7/202 | 15/200
Other Adverse Events (participants affected / at risk) | 94/834 | 32/202 | 23/202 | 25/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1 (N=834) | Etanercept 50 mg Plus MTX -Period 2 (N=202) | Etanercept 25 mg Plus MTX-Period 2 (N=202) | Placebo Plus MTX-Period 2 (N=200)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Refraction disorder (Eye disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Polyp colorectal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Cervicitis human papilloma virus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Psychiatric disorders (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Depression (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 Milligrams (mg) Plus Methotrexate (MTX)-Period 1 (N=834) | Etanercept 50 mg Plus MTX -Period 2 (N=202) | Etanercept 25 mg Plus MTX-Period 2 (N=202) | Placebo Plus MTX-Period 2 (N=200)
Nasopharyngitis (Infections and infestations) | 48 | 18 | 10 | 10
Bronchitis (Infections and infestations) | 0 | 12 | 11 | 6
Pharyngitis (Infections and infestations) | 0 | 3 | 5 | 11
Headache (Nervous system disorders) | 51 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.